CLINICAL TRIAL: NCT03360786
Title: Primary Prevention of Concussion in Youth Ice Hockey Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sport Injury Prevention Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Conc-PT-03
Record Dates: First submitted 2017-10-24; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Concussion
Keywords: sport concussion; cervical spine; youth
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An assessor who is blinded to group allocation will perform the pre and post assessment measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Protocol (Experimental): The intervention group will work with the study physiotherapist and perform a 10-20 minute progressive exercises twice per week. The intervention will include a series of exercises including dynamic balance, adaptation, cervical spine strength, cervical spine neuromotor control and divided attention exercises. Exercises will begin at a lower level and progress to increasingly difficult levels of each exercise type over the course of the intervention. Concussion education and injury identification will also be completed.
  Interventions: Other: Specific intervention
- Control Protocol (Active Comparator): The control group will continue with their standard warm up and practice schedule but have the addition of contact time with the study physiotherapist for education regarding concussion education and injury identification.
  Interventions: Other: Control intervention

INTERVENTIONS:
Other: Specific intervention — Series of progressive exercises targeted at balance, adaptation, dividing attention, head on neck control, visual + education on concussion identification and concussion education
  Arms: Specific Protocol
Other: Control intervention — Education on concussion and concussion identification in addition to typical cardiovascular warmups
  Arms: Control Protocol

SUMMARY:
1. Background and Rationale:

   Little is currently known about intrinsic risk factors for sport-related concussion in youth ice hockey players. Emerging research suggests that alterations in cervical and balance function increase the risk of concussion in youth ice hockey players. Thus, evaluation of a primary prevention program aimed at addressing alterations in cervical and vestibular function may result in a protective effect in reducing the risk of concussion. Such a program targeting intrinsic risk factors for concussion has not previously been evaluated and thus a pilot Randomized control trial (RCT) to inform the feasibility and efficacy of such a program is needed prior to proceeding to evaluation of such a program on a larger scale.
2. Research Question and Objectives

   The primary objectives of this pilot RCT study are: 1) To evaluate the feasibility of a concussion prevention program in youth ice hockey players; and 2) To evaluate the efficacy of a concussion prevention program in decreasing the risk of concussion. Exploratory objectives include evaluating the changes in quality of life, clinical measures of cervical and vestibular function measures and Hockey Canada on-ice skills testing in youth ice hockey players following a concussion prevention program.
3. Methods

This study will be a pilot RCT. Prior to the 2017 hockey season, 120 players from 8 youth ice hockey teams ages 13-17 will be recruited to participate. Once parental consent and/or player assent has been obtained, players will complete a series of initial intake forms. Baseline tests and measures, including a standardized preseason baseline questionnaire (regarding playing history, past medical history, participation in sport) and a battery of questionnaires and clinical measures. Individuals will be randomly allocated into either a control protocol (general cardiovascular warm-up, general stretching and strengthening, education on concussion identification) or a specific protocol (balance, neuromotor control, strength, vestibulo-ocular and oculomotor training + concussion education). Both groups will meet with the study physiotherapist once weekly for 4 weeks and exercises will be progressed. A previously validated prospective injury surveillance system will be implemented. As part of this process, a team designate will collect data throughout the season regarding individual player participation in games, practices and dry land training sessions. Individuals with a suspected concussion will be referred to the study sport medicine physician for evaluation, diagnosis and standard of care management. At this time all baseline tests and measures will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will broadly include individuals aged 13 - 17 years of age who are currently participating in organized ice hockey.

Exclusion Criteria:

* Inability to participate in physical activity for a reason other than sport related concussion.
* Inability to communicate in English language.
* Neurodevelopmental delays expected to affect ability to adapt with treatment.
* Orthopaedic or other injury affecting ability to participate.
* Medication known to affect neural adaptation as they may alter the response to treatment.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-29 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Concussion prevention protocol | 6 months (length of hockey season)
  A primary outcome of interest is diagnosis of concussion. This will be determined by the study sport medicine physician in accordance with current standards of care and as per the 5th International Consensus on Concussion in Sport Statement. Medical clearance to return to sport will be determined by the study sport medicine physician according to the 5th Consensus on Concussion in Sport Statement.
Number of participants able to complete protocol. | 6 months (length of hockey season)
  Number of participants completing each intervention will be calculated

SECONDARY OUTCOMES:
Pediatric Quality of Life Scale (PedsQL) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  The Pediatric Quality of Life Scale (PedsQL) is a measure of quality of life that is specific to children and measures four health domains including: Physical, emotional, social and school functioning. It is a measure that has demonstrated reliability and validity in multiple disease types in children, including traumatic brain injury. 0-100/100
Numeric Pain Rating Scale for Neck pain | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Neck pain rated from 0-10/10
Numeric Pain Rating Scale for Headache | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Headache pain rated from 0-10/10
Numeric Dizziness Rating Scale | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Dizziness rated from 0-10/10
Sport Concussion Assessment Tool 5 (SCAT5) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Multifaceted assessment tool including symptom reports (rated 0-6 for 22 different symptoms), Cognitive Screen (score /30), Neurological screen (Y/N for 5 questions and balance exam /30)
Dynamic Visual Acuity (DVA) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Clinical test of dynamic visual acuity using ETDRS chart
Head Thrust Test (HTT) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Clinical test to evaluate ability to maintain eyes on a stationary target. Performed to right and left. (+ve/-ve)
Functional Gait Assessment (FGA) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Dynamic balance measure including 10 different walking tasks that are rated on a scale of 0-3 for a total score out of 30
Advanced Functional Gait Assessment (A-FGA) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Newly created balance measure that represents a more difficult measure of dynamic balance and is a combination of progressively more difficult tasks included in the FGA. Clinician rated score 0-3 for each task. Total score out of 18
Walking While Talking Test (WWTT) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Test of walking and performing cognitive tasks of increasing difficulty, Time (seconds) for each task is recorded.
Cervical Flexion Endurance test (CFE) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Test performed in crook lying that measures the ability of a subject to maintain head in a craniovertebral flexion position and slightly lifted off pillow. Time (seconds)
Cervical Flexion Rotation Test (CFRT) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Screening test for upper cervical spine involvement. Positive/negative and is performed to both right and left.
Anterolateral cervical spine strength | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Measured using a head held dynamometer with subject in supine position. Test is repeated 3 times. Output measured in kg.
Head perturbation test (HPT) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  Ability to maintain head in a neutral position with external perturbation applied. Score out of 8 is recorded
Vestibular/Ocular Motor Screening Assessment (VOMS) | Time 0, 4 weeks, end of hockey season (approximately 6 months)
  As per Mucha et al, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Schneider, PT, PhD, Principal Investigator — Sport Injury Prevention Research Centre
Locations (1):
- University of Calgary Sport, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share individual participant data with others outside of the research team.